CLINICAL TRIAL: NCT03805061
Title: Evaluation of the Effects of Aerobic and Isokinetic Exercise Program on Muscle Power Cardiovascular System and Life Quality in Multiple Sclerosis Patients
Brief Title: Effects of Aerobic and Isokinetic Exercise in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sevgi Atar, Director of Administrative, Specialist, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 128
Record Dates: First submitted 2018-12-25; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; aerobic; isokinetic; exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 40 patients enrolled in the study from outpatient clinics were included. Two groups were formed, namely 'aerobic exercise' and 'isokinetic exercise' groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aerobic exercise group (Active Comparator): Group 1 was 'aerobic exercise group'. Patients in this group were included in an aerobic exercise rehabilitation program that they would apply for 3 days per week for 8 weeks. The aerobic exercise group by using treadmill their walking speeds were adjusted according to the maximum speed at which the person could walk was performed for a period of ; 8 weeks, 3 days a week, 30-45 minutes each patient according to the progressive exercise method. 5-10 minutes warm-up exercise was performed before starting to work, 5-10 minutes stretching exercise at the end of the exercise.
  Interventions: Other: 'aerobic exercise'
- Isokinetic exercise group (Active Comparator): Group 2 was 'isokinetic exercise group'. Patients in this group were included in an isokinetic exercise rehabilitation program that they would apply for 3 days per week for 8 weeks. Patients in the isokinetic exercise group pedaled a bicycle ergometer for warming with low resistance for 5 minutes before starting to exercise, and exercise was applied for 5-10 minutes to cool down at the end of the study.
  Interventions: Device: 'isokinetic exercise'

INTERVENTIONS:
Other: 'aerobic exercise' — The aerobic exercise group by using treadmill their walking speeds were adjusted according to the maximum speed at which the person could walk was performed a period of; 8 weeks, 3 days a week, 30-45 minutes each patient.
  Arms: Aerobic exercise group
Device: 'isokinetic exercise' — Patients in the isokinetic exercise group pedaled a bicycle ergometer for warming with low exercise and exercise was applied for 5-10 minutes to cool down at the end of the study. were included in a rehabilitation program that they would apply for 3 days per week for 8 weeks.The measuring of isokinetic muscle strength, CSMI Humac Norm isokinetic dynamometer's commonly used angular velocities of 60 ° and 180 ° / sec was used.
  Arms: Isokinetic exercise group

SUMMARY:
The investigators aimed in this study to measure the muscular strength, cardiovascular system and quality of life effects of rehabilitation with aerobic and isokinetic exercise program in MS patients.

DETAILED DESCRIPTION:
A total of 40 patients enrolled in the study from outpatient clinics were included. Two groups were formed, namely 'aerobic exercise' and 'isokinetic exercise' groups. Using modified Bruce protocol, effort capacities were measured with Humac Norm Cybex dynamometer, 6 min. walking distance and MSQOL-54 scale were used to assess the quality of life. The aerobic exercise group by using treadmill their walking speeds were adjusted according to the maximum speed at which the person could walk was performed for a period of ; 8 weeks, 3 days a week, 30-45 minutes each patient according to the progressive exercise method. 5-10 minutes warm-up exercise was performed before starting to work, 5-10 minutes stretching exercise at the end of the exercise. Patients in the isokinetic exercise group pedaled a bicycle ergometer for warming with low resistance for 5 minutes before starting to exercise, and exercise was applied for 5-10 minutes to cool down at the end of the study. The exercise program was applied for 8 weeks with 3 repetitions per week.

Assessment of exercise capacity (effort capacity) was performed by applying the Norav Trackmaster TMX 425 Treadmill Exercise Device by applying Modified Bruce protocol. Patients' total exercise times were expressed in seconds. Indirect maximum amount of oxygen volume (VO2 max) values were calculated using heart rate obtained with submaximal treadmill exercise.All the cases participating in the study were compared in terms of the pre-treatment MSQoL-54 scale and the MSQoL-54 scale subscale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multipl Sclerosis
* 18-65 years old adults
* Patients signed informed consent forms

Exclusion Criteria:

* Non-MS musculoskeletal system diseases
* Congenital anomalies, limb amputations
* Accompanying neurological diseases (Parkinson, Alzheimer, Polyneuropathy etc.)
* Vestibular system diseases
* Chronic diseases (diabetes mellitus, chronic obstructive pulmonary disease, hypertension, hyperlipidemia, severe cardiac disease, malignancy)
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04-30 (Actual); Primary Completion 2008-10-30 (Actual); Study Completion 2008-11-01 (Actual)

PRIMARY OUTCOMES:
Muscle strenght outcomes | 8 weeks
  The measuring of muscle strength, CSMI Humac Norm isokinetic dynamometer's commonly used angular velocities of 60 ° and 180 ° / sec was used. The muscle strenght peak torque value was newton-meter (Nm)
Quality of life outcomes | 8 weeks
  Quality of life was assesment via Multiple Sclerosis Quality of Life-54 instrument (MSQoL-54). MSQol-54 consists of 54 questions in total. In all cases, they were asked to fill in the questionnaire alone and by reading it themselves. The overall MSQoL-54 scale should be between in 0-100 scores. Higher scores better than lower scores.
The effort capacity outcomes | 8 weeks
  The effort capacity was performed by applying the Norav Trackmaster TMX 425 Treadmill Exercise Device by Applying Modified Bruce Protocol. The values of the effort capacity were assesment as maximum amount of oxygen volume (ml/kg/min.).

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Atar, M.D., Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization

IPD SHARING:
Plan to Share IPD: No
There is any plan to make IPD available to other researchers.